CLINICAL TRIAL: NCT06135922
Title: Multicenter, Open Label, Single-arm Exploratory Clinical Study of EBV-TCR-T Cells for EBV-associated Hemophagocytic Lymphohistiocytosis or EBV Infection
Brief Title: Clinical Study of EBV-TCR-T Cells for EBV-associated Hemophagocytic Lymphohistiocytosis or EBV Infection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2022-381-01
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: EBV-associated Hemophagocytic Lymphohistiocytosis; EBV Infection
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: EBV-TCR-T cells (Experimental): The patients with EBV-HLH or EBV infection will receive infusions of EBV-TCR-T cells, with the escalated dose ranging from 1×10^6/kg to 1×10^8/kg EBV-TCR-T cells per dose
  Interventions: Biological: EBV-TCR-T cells

INTERVENTIONS:
Biological: EBV-TCR-T cells — The patients with EBV-HLH or EBV infection will receive infusions of EBV-TCR-T cells, with the escalated dose ranging from 1×10^6/kg to 1×10^8/kg EBV-TCR-T cells per dose.

SUMMARY:
This is a multi-center, single arm, open-label, phase I study to determine the safety and effectiveness of EBV-TCR-T cell immunotherapy in treating EBV-associated hemophagocytic lymphohistiocytosis (EBV-HLH) or EBV infection

DETAILED DESCRIPTION:
Epstein-Barr virus (EBV) is a widely disseminated herpesvirus that is spread by intimate contact between susceptible persons and asymptomatic EBV shedders. The inability to control EBV infection can lead to some patients developing EBV-positive B-cell lymphomas, chronic active EBV infections, and hemophagocytic lymphohistiocytosis (HLH). In this prospective study, HLA-A*02:01/11:01/24:02-restricted EBV-specific T cell receptor (TCR) will be introduced into the T cells of donors by ex vivo lentiviral transduction to generate EBV-TCR-T cells. An escalated dose ranging from 1×10^6/kg to 1×10^8/kg of EBV-TCR-T cells will be infused into patients with EBV-HLH or EBV infection. The safety, efficacy, pharmacokinetics and cytokine levels of allogenic EBV-TCR-T cell therapy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-60 years, gender unlimited.
* Diagnosed with EBV associated-hemophagocytic lymphohistiocytosis (HLH) or EBV infection.
* Fully understood and informed the study and signed the ICF.
* Karnofsky Score ≥ 70(age ≥16y) or Lansky Score ≥ 50(age<16y).
* TCRT-T cell donor inclusion criteria: 1)Age >=8 years, gender unlimited; 2) Understand and voluntarily sign informed consent and are willing to comply with laboratory tests and other research procedures; 3) ≥ 3/6 HLA match with TCR-T cell recipients enrolled; 4) Lymphocyte count = (0.8~4) × 10^9/L; 5) Have sufficient venous circulation, without any symptoms that do not allow blood cell isolation.

Exclusion Criteria:

* Patients with uncontrolled active aGVHD one day before TCR-T cell infusion.
* Patients with severe kidney disease (Cr > 3×normal value), liver damage (TBIL >2.5×upper limit of normal value, ALT and AST > 3×upper limit of normal value) or heart failure (NYHA heart function grade IV or left ventricular ejection fraction<50%) one week before TCR-T cell infusion.
* Anticipated to take immunosuppressive hormones on the day of TCR-T cell infusion.
* Use of immunosuppressive drugs or G-CSF within 2 weeks before PBMC blood collection.
* Have tumours, active and uncontrolled malignant diseases.
* Serologically positive for HIV-Ab or TAP-ab.
* Pregnant or lactating women.
* Men and their partners or women of childbearing potential refused contraception during the study period.
* Anticipated to have other cell therapies in 4 week post TCR-T cell infusion.
* Participated in any other clinical study of drugs and medical devices before 4 weeks of enrollment.
* Allergy to albumin.
* TCRT-T cell donor exclusion criteria: 1) pregnant woman; 2) Serologically positive for HBsAg, HCV-Ab, HIV-Ab or TAP-ab; 3) EBV-DNA or CMV-DNA positive; 4) other uncontrolled infection; 5) Use of immunosuppressive drugs or G-CSF within 2 weeks before PBMC blood collection.

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year after EBV-TCR-T treatment
  Percentage of participants with adverse events

SECONDARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days after EBV-TCR-T treatment
  Toxic effects considered by the investigators to be related to the EBV-TCR-T
Maximum tolerated dose （MTD） | 28 days after EBV-TCR-T treatment
  The highest dose of DLT was seen in 1/6 of subjects
The proportion of EBV-DNA negative patients | 180 days after EBV-TCR-T treatment
  The proportion of patients EBV-DNA negative after EBV-TCR-T treatment
The time to EBV-DNA negative | 180 days after EBV-TCR-T treatment
  The time from the start of therapy to EBV-DNA negative detected
Changes of EBV-DNA copies number | 1 year after EBV-TCR-T treatment
  Quantitative PCR will be used to determine viral copy numbers in peripheral blood.
Maximum Plasma Concentration (Cmax) of EBV-TCR-T cells | 28 days after EBV-TCR-T treatment
  Cmax of EBV-TCR-T cells in patients with EBV-HLH or EBV infection
Area under the plasma concentration versus time curve (AUC) of EBV-TCR-T cells | 28 days after EBV-TCR-T treatment
  AUC of EBV-TCR-T cells in patients with EBV-HLH or EBV infection
Time to peak (Tmax) of EBV-TCR-T cells | 28 days after EBV-TCR-T treatment
  Tmax of EBV-TCR-T cells in patients with EBV-HLH or EBV infection
Half life time (T1/2) of EBV-TCR-T cells | 28 days after EBV-TCR-T treatment
  T1/2 of EBV-TCR-T cells in patients with EBV-HLH or EBV infection

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China